CLINICAL TRIAL: NCT04507217
Title: A Phase II, Open-Label, Multicenter, Prospective Clinical Study to Investigate the Efficacy and Safety of Tislelizumab Combined With Pemetrexed/ Carboplatin in Patients With Brain Metastases of Non-squamous Non-small Cell Lung Cancer
Brief Title: Tislelizumab Combined With Pemetrexed/ Carboplatin in Patients With Brain Metastases of Non-squamous NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2003-IIT
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: NSCLC Stage IV; Brain Metastases; PD-1 Antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — tislelizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Tislelizumab Combined with Pemetrexed/ Carboplatin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients (Experimental): tislelizumab (200mg) in combination with pemetrexed (500mg/m2) and carboplatin (AUC=5) intravenously on day 1 of a 3-week cycle for 4 cycles. Afterwards, patients without disease progression were treated with maintenance treatment with tislelizumab (200mg) plus pemetrexed (500mg/m2) every 3 weeks up to 24 months or until disease progression, unacceptable toxicity, or death.
  Interventions: Drug: Tislelizumab, Carboplatin, Pemetrexed

INTERVENTIONS:
Drug: Tislelizumab, Carboplatin, Pemetrexed — Tislelizumab: 200mg administered intravenously (IV) on Day 1 of each 21-day cycle
  Carboplatin: AUC 5 administered intravenously (IV) on Day 1 of each 21-day cycle, 4 cycles
  Pemetrexed: 500mg/m2 administered intravenously (IV) on Day 1 of each 21-day cycle

SUMMARY:
This is a phase II, Open-Label, Multicenter, Prospective Clinical Study to Investigate the Efficacy and Safety of Tislelizumab Combined with Pemetrexed/ Carboplatin in Patients with Brain Metastases of Non-squamous Non-small Cell Lung Cancer. The primary end point is PFS, and secondary endpoint is ORR, OS, DoR and Neurocognitive impairment. during the study, the exploratory objectives including (1) PD-L1 expression, TMB, and other potential predictive biomarkers, correlated with response to treatment (2) Progression-free survival based on intracranial response (iPFS) according to RECIST 1.1 and RANO-BM

ELIGIBILITY:
Inclusion Criteria:

Disease-related inclusion criteria:

1. Histologically confirmed metastatic (Stage IV) not amenable to curative surgery or radiotherapy, non-squamous NSCLC according to American Joint Committee on Cancer (AJCC), 8th Edition.
2. Radiographically confirmed brain metastases;
3. No prior systemic treatment for stage IV NSCLC. (Bevacizumab administered for improving radiation-induced encephaledema during irradiating intracranial lesions is not considered as systemic therapy for stage IV NSCLC)
4. Patients with asymptomatic BM or symptoms can be controlled by low dose corticosteroids (≤ 10 mg/day of prednisone or equivalent) or antiepileptics drugs;
5. Patients with previous local treatment to BMs should be stable and suitable to receive the systemic treatment;
6. ECOG PS: 0 ~ 1
7. Extracranial measurable target lesions (per RECIST v1.1)
8. Life expectancy ≥ 3 months

   Have adequate hematology, clinical chemistry, and organ function as indicated by the following laboratory values (confirmed within 7 days prior to the first dose):
9. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 90 g/L.
10. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × upper limit of normal [ULN].
11. Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
12. Serum total bilirubin ≤ 1.5 × ULN (total bilirubin must be < 3 × ULN for patients with Gilbert's syndrome).
13. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN or AST and ALT ≤ 5 × ULN for patients with liver metastases.

    General inclusion criteria:
14. Able to provide written ICF signed by patient or by his/her legally authorized representative or guardian and can understand and agree to comply with the study protocol and follow-up procedures.
15. Male or female, aged 18 ~ 75 years on the day of signing ICF. Female patients of childbearing potential and non-sterile male patients must be willing to use a highly effective method of birth control for the duration of the study and for at least 120 days after the last dose of tislelizumab.

Exclusion Criteria:

Disease-related exclusion criteria:

1. Received prior therapies targeting PD-1, PD-L1, CTLA-4 or other immune checkpoints inhibitors.
2. Received prior systemic chemotherapy for advanced disease.
3. Have EGFR mutation or ALK gene translocation.
4. Patients iwith BMs that have received systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent) or other drugs to relieve or prevent symptoms of BMs.
5. Patients with intracranial metastases that are locally amenable.
6. Have received any approved systemic anticancer therapy or systemic immunomodulators (including but not limited to interferon, interleukin-2, and tumor necrosis factor) within 4 weeks prior to the first dose of study drug.
7. Have clinically uncontrolled pleural effusion or ascites that requires pleurocentesis or abdominal tapping for drainage within 2 weeks prior to the first dose of study drugs.
8. Active leptomeningeal metastasis.

   Exclusion criteria related to study drugs:
9. History of allergic reactions to any study drugs and their excipients.
10. Creatinine clearance (Ccr) < 45 mL/min.
11. Patients with active viral hepatitis that requires treatment as judged by the investigator: a. chronic hepatitis B virus carriers with HBV DNA ≥ 500 IU/mL (2500 copies/mL) (The HBV DNA test will be performed only for patients who have a positive antibody to hepatitis B core antigen (anti-HBc antibody) test); b. patients who have positive hepatitis C virus (HCV) RNA results (The HCV RNA test will be performed only for patients testing positive for HCV antibody).
12. Active autoimmune diseases that requires systemic treatment and may impact study treatment as assessed by investigator.
13. Any condition that required extensive chronic treatment with either corticosteroids or any other immunosuppressive medications that may impact study treatment as assessed by investigator.

    General exclusion criteria:
14. Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral therapy, including tuberculosis infection, etc.; 1) Serious infections within 4 weeks before first dose, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia; 2) Receive therapeutic oral or intravenous antibiotics within 2 weeks before first dose. With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung diseases, etc.
15. Major surgery requiring general anesthesia within 4 weeks before first dose.
16. Underlying medical conditions or alcohol or drug abuse or dependence that are to be unfavorable for the administration of study drugs or may have affected the interpretation of the results or rendered the patient at high risk from treatment complications.
17. Concurrent participation in another therapeutic clinical study. Female patients who are pregnant, breastfeeding, or males and females patients planning to have child during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) rate at 12 months according to RECIST v1.1 | 12months
  Progression-free survival is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST v1.1 | 36 months
  ORR is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR).
Progression-free survival (PFS) according to RECIST v1.1 | 12 months
  Progression-free survival is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first.
Overall Survival (OS) | 36 months
  OS is defined as the time from the starting date of study drug to the date of death due to any cause
Progression-free survival (PFS) according to RANO-BM | 36 months
  PFS2 is defined as the time from first intracranial disease progression to second/subsequent disease progression (intracranial or extracranial) after initiation of new anti-cancer therapy, or death from any cause, whichever occurs first
Duration of Response (DoR) according to RECIST v1.1 | 36 months
  DoR is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first
Incidence and severity of treatment-emergent AEs (TEAEs) | 36 months
  TEAEs graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Neurocognitive impairment | 36 months
  Neurocognitive impairment according to Hopkins Verbal Learning Test-Revised（HVLT-R）

OTHER OUTCOMES:
PD-L1 expression, TMB, and other potential predictive biomarkers, correlated with response to treatment | 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning